CLINICAL TRIAL: NCT00487578
Title: Evaluation of the Efficacy of Naratriptan for the Treatment and Prevention of Post Traumatic Headache Associated With Cognitive Dysfunction
Brief Title: Naratriptan for the Treatment of Post Traumatic Headache Associated With Cognitive Dysfunction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated October 2009 (in 4th year) due to low enrollment and anticipated drug expiration November 2009.
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry); Clinvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106542
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Post Traumatic Headache
Keywords: Post traumatic headache; Head trauma; Head injury; Headache; Naratriptan
MeSH Terms: conditions — Post-Traumatic Headache; Craniocerebral Trauma; Headache | interventions — naratriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Naratriptan 2.5 mg tablet bid x 30 days
  Interventions: Drug: naratriptan HCl
- B (Placebo Comparator): placebo matching naratriptan 2.5 mg tablet
  Interventions: Drug: naratriptan HCl

INTERVENTIONS:
Drug: naratriptan HCl — naratriptan 2.5mg tablet bid x 30 days OR matching placebo
  Other Names: Amerge

SUMMARY:
The purpose of this study is to determine whether naratriptan, a medication approved for treatment of migraine, is effective in the treatment of post traumatic headache associated with cognitive dysfunction.

DETAILED DESCRIPTION:
Naratriptan has demonstrated efficacy in relieving headache. Other studies have demonstrated that primary headaches with at least one headache feature are likely to respond to triptans. In addition, there are anecdotal reports of triptans being effective in post traumatic headaches, especially if headache features are noted in the patient's history. Further, there are several small pilot studies with triptans demonstrating a prompt improvement in headache-induced cognitive changes. Cognitive performance can be measured by the Mental Efficiency Workload Test (MEWT), a handheld Palm neuropsychological test battery that measures mental efficiency. This tool can be used to demonstrate short and long term improvement in mental status beyond that seen at baseline.

Informal observations by the protocol authors have suggested that the use of triptans on a routine basis may ameliorate the headache and associated symptomatology of post traumatic headache. Therefore, this study is undertaken to study the use of naratriptan in the treatment of post traumatic headache. Roger K. Cady, MD, serves as the sponsor. The study is funded by GlaxoSmithKline.

56 subjects with a formal diagnosis of Chronic post-traumatic headache attributed to mild head injury (IHS/ICHD-II 5.2.2) and with self-reported mild cognitive inefficiency secondary to headache will be enrolled. Subjects meeting inclusion criteria will complete a physical examination and baseline testing and be randomized 1:1 to naratriptan 2.5mg bid x 30 days or a matched placebo bid x 30 days. A daily diary will document response to treatment. Subjects will return to the clinic at Day 10 and Day 30 and complete phone contacts at Days 5, 15, 21, 32 and 90. Information will be collected throughout the study on questionnaires related to headache impact, general health, satisfaction with medication, and quality of life. Cognition will be measured using the MEWT.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-55. A female is eligible to enter and participate if she is of: non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or, child-bearing potential, has a negative pregnancy test (urine or serum) at screen, and agrees to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study; subjects utilizing this method must agree to use alternate method of contraception if they become sexually active and will be queried on whether they have been abstinent when they present to the clinic for the Final Visit or, Female sterilization; or, Sterilization of male partner; or, Implants of levonorgestrel; or, Injectable progestogen; or, Oral contraceptive (combined or progestogen only); or, Any intrauterine device (IUD) with published data showing highest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or, Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm). Any other barrier methods (only if used in combination with any of the above acceptable methods) or, Any other methods with published data showing highest expected failure rate for that method is less than 1% per year.
* Formally diagnosed ICHD 5.2.2 chronic post traumatic headache
* Have had traumatic brain injury (TBI) not more than 5 years prior to enrollment
* Medically stable as determined by Investigator
* On stabilized dosage of any headache preventive medications for 3 months prior to screening
* On stabilized dosage of concomitant medications at discretion of investigator
* Chronic headache history only after the TBI
* Able to understand and communicate intelligibly with study observer
* Able to take oral medication, adhere to the medication regimens and perform study procedures
* Able to read and comprehend written instructions and be willing to complete all procedures and assessments required by protocol
* Subject is able to demonstrate willingness to participate by signing and understanding an informed consent after full explanation of study
* Self-reported cognitive inefficiency or "brain-fog" during headache

Exclusion Criteria:

* History of hypersensitivity to triptan-like medication
* Pathology of salivary glands such as sialadenitis (e.g., Sjorgen's Syndrome, viral or bacterial sialadenitis, or obstructive sialadenitis)
* Any condition or symptom that would knowingly alter content of saliva
* History of, symptoms or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes or other significant underlying cardiovascular disease. Ischemic cardiac syndromes include, but are not limited to, angina pectoris of any type (e.g. stable angina of effort and vasospastic forms of angina such as Prinzmetal variant, all forms of myocardial infarction, and silent myocardial ischemia. Cerebrovascular syndromes include, but are not limited to, strokes of any type as well as transient ischemic attacks. Peripheral vascular disease includes, but is not limited to, ischemic bowel disease.
* Any medication overuse that in the opinion of the investigator has exacerbated or contributed to current headache pattern of subject
* Uncontrolled hypertension, severe renal impairment, severe hepatic impairment, hemiplegic or basilar headache
* History of hypersensitivity to naratriptan or any components
* Pregnant, trying to get pregnant, or lactating
* Recent history of abuse of alcohol or other drugs that would interfere with participation
* Participation in another investigative drug study within previous 30 days
* Chronic pain syndromes, fibromyalgia, Gulf War Syndrome, and other multisystem diseases characterized by poor or no response to pain-reducing interventions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (3):
- United States (3):
  - Clinvest, Springfield, Missouri
  - Carolinas Rehabilitation, Carolinas HealthCare System, Charlotte, North Carolina
  - Anodyne Headache and Pain Care, Dallas, Texas

REFERENCES:
- [Background] Baandrup L, Jensen R. Chronic post-traumatic headache--a clinical analysis in relation to the International Headache Classification 2nd Edition. Cephalalgia. 2005 Feb;25(2):132-8. doi: 10.1111/j.1468-2982.2004.00818.x. PMID 15658950
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment started in 2006 at Site 1 (headache specialty clinic). Subjects were never enrolled at 2nd site (hospital rehabilitation center). Sites 3 (pain clinic) and 4 (hospital rehabilitation center) were added in 2008. Enrollment continued until study termination October 2009.
Pre-assignment Details: 19 participants were screened. 7 were Screen Failures.
Groups:
- Active Naratriptan: Naratriptan 2.5 mg tablet twice daily (bid) x 30 days
- Placebo Matching Naratriptan: placebo matching naratriptan 2.5 mg tablet twice daily (bid) x 30 days
Period: Overall Study
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Started | 3 | 9
Completed | 2 | 5
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan | Total
Number analyzed (Participants) | 3 | 9 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 12
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.66 (10.96) | 37.22 (9.65) | 37.83 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: Number of headache days as measured by the Headache Diary
Time Frame: Day 30
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Headache Impact Test-6 (HIT-6) Score
Description: Impact of headache symptoms on subject's life as measured by HIT-6 questionnaire scores. Possible scores range from 36 to 78. Score of 48 or less indicates headache has little impact on life. Score of 60-78 indicative of very severe impact.
Time Frame: Day 0, Day 30
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Mental Efficiency Workload Test (MEWT) Performance Index Score
Description: Cognitive function as measured by Performance Index scores on the Mental Efficiency Workload Test (MEWT). On the performance index scale of 1 to 10, 1 indicates the poorest level and 10 indicates the best level of cognitive functioning. Tests include: Simple reaction time, Running memory, Matching to sample, Math processing and a sleep scale.
Time Frame: Day 0, Day 10, Day 30
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Satisfaction With Medication Score
Description: Subject overall satisfaction with effectiveness of the therapy as measured by score on the Satisfaction with Medication questionnaire. Scale range: Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied.
Time Frame: Day 30, Day 90
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life Scores
Description: Quality of life as measured by Migraine Specific Quality of Life questionnaire (MSQ) scores. 14 questions ask how often headaches have interfered with specific daily activities in previous 4 weeks. 6-point scale ranges from "None of the time" to "All of the time".
Time Frame: Day 0, Day 30, Day 90
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sustained Treatment Effect
Description: Sustained treatment effect as measured by the MEWT Performance Index score compared to change in number of Headache Days. Results would be presented in the form of a correlation analysis. There is an expected negative correlation as performance index increases and number of headache days decrease (a correlation of -1).
Time Frame: Day 0, Day 10, Day 30
Population: No analysis was conducted. Study terminated due to expiration of study medication and low enrollment.
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Description: AEs collected from Diaries reviewed at Visit 2/Day 10 and Visit 3/Day 30. AEs collected during phone interviews (Days 5, 15, 21, 32, and 90).
Arm/Group | Active Naratriptan | Placebo Matching Naratriptan
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Naratriptan (N=3) | Placebo Matching Naratriptan (N=9)
nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Drowsiness (Renal and urinary disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased headache severity (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Change in headache location (Nervous system disorders) | 0 (0) | 1 (1)
Change in headache sensation (Nervous system disorders) | 0 (0) | 1 (1)
Achiness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2) — Referred to cardiologist. Stress ECG performed. All normal. Pt unblinded.
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Stomach tenderness (General disorders) | 0 (0) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Twitching eye (General disorders) | 0 (0) | 1 (1)
Increased twitching left arm (General disorders) | 1 (1) | 0 (0)
Increased headache frequency (Nervous system disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Itching neck (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itching eyes (General disorders) | 0 (0) | 1 (1)
Redness of face (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Feels hot and cold (General disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Unbalanced gait (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated October 2009 (in 4th year) due to low enrollment and anticipated drug expiration November 2009 (study drug had previously been re-supplied at expiration of 1st batch November 2007).

No analysis performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study data collected by Investigator is authorized subject to the following:Investigator is free to publish results of its part of study in collaboration with other investigators subsequent to the multicenter publication issued by Clinvest. If no multicenter publication is submitted within 12 months of end of study, investigator may publish results of its data. Investigator shall submit a copy of manuscript or abstract to Clinvest for review 30 days prior to journal submission.